CLINICAL TRIAL: NCT06721299
Title: Clenbuterol to Target DUX4 in FSHD (Target FSHD): Open Label Safety and Tolerability Study of 3 Doses of Clenbuterol
Brief Title: Clenbuterol to Target DUX4 in FSHD
Acronym: Target FSHD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey Statland (Other)
Collaborators: University of Washington (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of Rochester (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Statland, Professor of Neurology, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00150777; P50AR065139 (NIH)
Record Dates: First submitted 2024-09-05; First posted 2024-12-06 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Muscular Dystrophy, Facioscapulohumeral
Keywords: FSHD
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral | interventions — Clenbuterol

STUDY DESIGN:
Intervention Model Description: Three sequential multiple ascending dose cohorts (of n=10 participants)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Clenbuterol Cohort 1 (Experimental): 20 mcg taken orally twice daily
  Interventions: Drug: Clenbuterol
- Clenbuterol Cohort 2 (Experimental): 40 mcg taken orally twice daily
  Interventions: Drug: Clenbuterol
- Clenbuterol Cohort 3 (Experimental): 60 mcg taken orally twice daily
  Interventions: Drug: Clenbuterol

INTERVENTIONS:
Drug: Clenbuterol — Beta-Agonist

SUMMARY:
The purpose of this study is to determine if Clenbuterol is a therapeutic option for FSHD by determining the safety and tolerability of the medication at three different dose levels.

DETAILED DESCRIPTION:
Clenbuterol is an EMA approved drug for COPD that three independent patient derived screens identified as suppressing DUX4 expression in cultured FSHD muscle. Prior clinical studies with related beta2-agonists showed some activity in FSHD but did not meet their primary endpoint, although the prior studies would likely have been designed differently with current knowledge. Target FSHD is a 6-month open-label multiple ascending dose study of clenbuterol for safety and tolerability to determine the best dose for a future trial of efficacy. In addition, this study will collect secondary outcome data on muscle function, MRI changes (lean muscle volume, fat infiltration, STIR-rating) and molecular markers of disease activity (histopathology and pre-determined baskets of DUX4-target, inflammation, and ECM genes) at the beginning and end of the study to assess and power their utility as measures of drug activity in a future interventional study of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of FSHD type 1 or 2, or have a clinical diagnosis of FSHD type 1 with a first degree relative with confirmed mutation
* between 18 and 75 years of age
* with a clinical severity score between 1 and 4
* Able to walk 30ft without support of another person
* Showing anti-gravity strength on at least one of the tibialis anterior muscles or having an MRI eligible muscle in the leg for needle biopsy
* willing and able to provide informed consent

Exclusion Criteria:

* Pregnant or planning to become pregnant during the conduct of the study
* have a poorly controlled medical condition
* Were involved in a study of an experimental agent within 3 months of enrollment
* Are taking beta-blockers or anabolic agent or potassium wasting diuretics
* have any condition or contraindication which would interfere with testing or preclude use of beta-agonist
* Are taking blood thinners or medications which make a needle muscle biopsy contra-indicated
* Are taking any medications or therapies with a contraindication to Clenbuterol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of Clenbuterol-related adverse reactions | from baseline to 6 month visit
  Patient report and medical records will be used to document adverse events and severe adverse events. Adverse events and severe adverse events will be assessed by the investigator and reported as needed for safety.
change in heart rate | from Month 1 to Month 6 visit
  Review of Vitals
change in blood pressure | from Month 1 to Month 6 visit
  Review of Vitals
Safety Lab Potassium (K) | Baseline to month 6 visit
  patient safety measured by potassium for signs of hypokalemia
Safety Lab Glucose | Baseline to month 6 visit
  Patient safety measured by blood glucose abnormalities
Tolerability of 3 doses of clenbuterol in sequential cohorts | from baseline to 6 month visit
  Tolerability will be defined as completing an arm without any clenbuterol related adverse events causing someone to withdraw
Safety ECG | from Month 1 to Month 6 visit
  Looking for sympathomimetic side effects such as cardiac arrhythmias
Safety Lab Creatine kinase (CK) | Baseline to Month 6 visit
  Patient Safety measured by creatine kinase abnormalities

SECONDARY OUTCOMES:
MRI | Screening to Month 6 Visit
  MRI measurements are considered gold standard for lean muscle volume measurement and disease biomarkers (fat volumes, fat faction, and STIR+ presence) that may be modulated by treatment. In addition, we will include analysis to help make needle biopsy based on STIR and quantitative fat fraction more efficient with higher yield using standard fiducial markings and body landmarks.
Muscle Biopsy for RNA sequencing | Baseline and Month 6
  change in a set of DUX4-regulated genes as measured in muscle using RNA sequencing. goal is to better understand the molecular changes in muscle tissue effected by the use of Clenbuterol.
FSHD-COM | Screening to Month 6 Visit
  An 18-item evaluator administered instrument comprised of individually validated functional motor task.the body regions assessed match areas of importance identified by patients and include leg function; shoulder and arm function; trunk function, hand function; and functional balance
Manual Muscle Testing (MMT) | Screening to Month 6 Visit
  a modified Medical Research Council 13-point scale with standardized positions for each muscle will help look at subject's change in strength over time.
Quantitative Muscle Testing (QMT) | Screening to Month 6 Visit
  Will test 5 bilateral muscles using a fixed myometry testing system with a force transducer attached by an inelastic strap to a metal frame, This will help us assess subjects change in strength
Patient Reported Outcome Measurement Information System-57 (Promis57) | Screening to Month 6 Visit
  The PROMIS57 is an instrument developed by the NIH which generates scores for physical function, and the impact of physical limitations on daily life. 57 questions are summed into a total score, which is transformed into a normalized t-score with 50 representing normal, and lower scores representing increasing disability.
FSHD Rasch-built overall disability scale (FSHD-RODS) | Screening to Month 6 Visit
  The FSHD-RODS is a questionnaire about the relationship between daily activities and health. 32 questions are are constructed using a modern clinimetric technique, the Rasch analysis, which by ordering the items in increasing difficulty, allows for the calculation of the sum of item scores to achieve a total score. Answers provide information about how FSHD affects daily and social activities and to what degree participants are able to perform usual activities.
Upper Extremity Functional Index (UEFI) | Screening to Month 6 visit
  This index measures upper extremity dysfunction. 20 questions are combined into a total score, the score is transformed into a normalized score with 80 representing normal, and lower scores representing increasing disability.
Clinical Global Impression of Severity and Change (CGI-S and CGI-C) | Screening to Month 6 visit
  Is a rating scale that measures symptom severity and change in severity in response to treatment in clinical trials.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Rochester Medical Center, Rochester, New York
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No